CLINICAL TRIAL: NCT06922890
Title: A Single-center, Prospective Investigator-initiated Trial to Evaluate the Safety and Exploratory Efficacy of STUP-001 in Patients With Chronic Spinal Cord Injury of AIS-A or B Level
Brief Title: First-in-Human Clinical Trial of STUP-001, an In Vivo Direct Cell Conversion Gene Therapy for AIS-A/B Chronic Spinal Cord Injury
Acronym: STUP-001
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: Stand Up Therapeutics INC. (Industry)
Responsible Party: Principal Investigator, Yoon Ha, Professor, Department of Neurosurgery, M.D., Ph.D., Yonsei University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUP-001_PRT; Stand Up Tx1 (Other: Stand Up Therapeutics, Inc.)
Record Dates: First submitted 2025-04-03; First posted 2025-04-11 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Spinal Cord Injury; Chronic Spinal Cord Injury
Keywords: Direct Lineage Reprogramming; Cell Fate Conversion; First-in-Human Multi-Cistronic Vector Application
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STUP-001 (1/2X) (Experimental): The participant with chronic spinal cord injury was administered a total of 25 μL via the intraparenchymal route into the spinal cord.
  Interventions: Drug: STUP-001
- STUP-001(1X) (Experimental): The participant with chronic spinal cord injury was administered a total of 50 μL via the intraparenchymal route into the spinal cord.
  Interventions: Drug: STUP-001

INTERVENTIONS:
Drug: STUP-001 — in vivo direct cell conversion gene therapy investigational product

SUMMARY:
This study aim to investigate the safety and exploratory efficacy of STUP-001 which is AAV-based spinal cord injury investigational product.

DETAILED DESCRIPTION:
Traumatic spinal cord injury (tSCI) often leads to irreversible paralysis and severely diminishes quality of life. Despite its profound impact, no fundamental treatment is currently available.

STUP-001, developed by Stand Up Therapeutics, Inc. under the leadership of Dr. Junsang Yoo, is an investigational in vivo gene therapy designed to directly convert astrocytes into functional neurons within the spinal cord. In preclinical studies, STUP-001 demonstrated both successful astrocyte-to-neuron conversion and meaningful improvements in motor function.

Building on these findings, this single-center, prospective, investigator-initiated clinical trial - "A Single-center, Prospective, Investigator-Initiated Trial to Evaluate the Safety and Exploratory Efficacy of STUP-001 in Patients with Chronic Spinal Cord Injury of AIS-A or B Level" - aims to assess the safety and exploratory efficacy of STUP-001 in patients aged 19 to 60 years with chronic SCI classified as AIS-A or B. Including the screening phase, each participant will undergo a 7-month evaluation period, during which safety, tolerability, and preliminary efficacy endpoints will be closely monitored.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged 19 to 60 years at the time of obtaining informed consent.
* Patients diagnosed with traumatic spinal cord injury classified as ASIA Impairment Scale (AIS) grade A or B:

  1. AIS-A: Complete loss of sensory and motor function.
  2. AIS-B: Partial preservation of sensory function with complete motor paralysis
* Patients who have been diagnosed with traumatic spinal cord injury for at least 6 months at the time of screening.

At the time of screening, women must provide evidence of non-fertile status by meeting at least one of the following criteria:

(a) Postmenopausal women: Defined as women over the age of 50 who have been amenorrheic for at least 12 consecutive months after discontinuing all exogenous hormonal treatments.

(b) Women with irreversible surgical infertility, including hysterectomy, bilateral oophorectomy, or bilateral salpingectomy. (Tubal ligation is not accepted.) (c) Women 50 years or younger who have been amenorrheic for at least 12 consecutive months after discontinuing all exogenous hormonal treatments and have luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels within the postmenopausal range defined by the study site.

* Acceptable methods of contraception include:

  1. Complete abstinence.
  2. Tubal sterilization.
  3. Hormonal contraceptives with no known drug interactions (e.g., levonorgestrel intrauterine system (IUS) (Mirena), medroxyprogesterone).
  4. Copper intrauterine device (IUD).
  5. Partner vasectomy. (Note: Periodic abstinence methods (e.g., ovulation timing, symptothermal method, or post-ovulatory methods) and withdrawal are NOT considered acceptable contraception methods.)
* Individuals who are able to understand the provided information and can voluntarily sign the written informed consent (or have a legally authorized representative sign on their behalf).

Exclusion Criteria:

* Patients diagnosed with traumatic spinal cord injury (SCI) classified as AIS-C or D at the time of screening.
* Patients with the following cardiovascular conditions at the time of screening:

  1. Myocardial infarction or unstable angina within the past 6 months.
  2. QTc interval ≥ 450 msec or clinically significant electrocardiographic (ECG) abnormalities.
  3. Congestive heart failure (CHF) classified as New York Heart Association (NYHA) Class II or higher.
  4. Stroke or transient ischemic attack (TIA) within the past 6 months.
* Patients with uncontrolled diabetes mellitus (e.g., HbA1c > 8% at screening).
* Patients with uncontrolled hypertension (e.g., systolic BP > 180 mmHg or diastolic BP > 100 mmHg).
* Patients diagnosed with, undergoing treatment for, or with a history of malignancy within the past 5 years at the time of screening.
* Patients with positive serologic test results for HBsAg, anti-HCV Ab, or anti-HIV Ab at the time of screening. However, patients with positive anti-HCV Ab may be eligible if HCV RNA test results are negative after treatment.
* Patients with clinically significant severe infections, as determined by the investigator (e.g., infections requiring continuous concomitant medication for ≥3 weeks during the clinical trial period).
* Patients with a history of hypersensitivity to any component of the investigational drug.
* Patients with a history of gene or cell therapy involving AAV2.
* Patients with the following abnormal laboratory test results at screening:

  1. WBC < 2,000/mm³
  2. Platelet count < 100,000/mm³
  3. Hemoglobin < 10.0 g/dL
  4. Serum creatinine > 1.5×ULN
  5. Total bilirubin > 1.5×ULN
  6. AST, ALT > 3×ULN
  7. PT-INR/aPTT > 1.5×ULN
* Patients with substance abuse, alcohol dependence, or psychiatric disorders.
* Patients who are unable to undergo general anesthesia.
* Pregnant or breastfeeding women, or those with a positive pregnancy test at screening.
* Patients who have received another investigational drug within 4 weeks prior to screening. However, patients who have not received an investigational drug or participated in non-interventional observational studies may be eligible.
* Any other individuals deemed ineligible for the clinical trial at the investigator's discretion.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dos-limit toxicity evaluation post STUP-001 administration | 4weeks post STUP-001 administration
  National Cancer Institute-Comone Terminology Criteria for Adverse Events V5.0 (NCI-CTCAE V5.0)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No